CLINICAL TRIAL: NCT05075317
Title: Time Restricted Eating and Cardiac Rehabilitation
Acronym: TREat-CR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-5510
Record Dates: First submitted 2021-06-16; First posted 2021-10-12 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
Keywords: Time-Restricted Eating; Cardiac Rehabilitation; Cardiorespiratory Fitness; Caloric Restriction; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard cardiac rehabilitation (Active Comparator): The 16-week program consists of physician-directed risk factor management, an individualized aerobic and resistance exercise prescription, and virtual education on disease management and lifestyle behaviors (including exercise safety, stress management, and heart-healthy nutrition), and an assessment with a registered dietitian and individualized recommendations for a heart-healthy diet. Additionally, selected patients with identified issues such as depression, anxiety, trouble sleeping, anger and social and emotional issues will receive one-on-one counselling with a psychologist or social worker.
  Interventions: Behavioral: Standard cardiac rehabilitation
- Standard cardiac rehabilitation + TRE (Experimental): Participants in this group will receive the same standard assessment and individualized recommendations as the comparator group, but will also be counselled to restrict their eating to between 11 am and 7 pm during the program starting the evening of the consultation. They will also be advised to perform their home-based exercise sessions during the fasting period in the morning.
  Interventions: Behavioral: Standard cardiac rehabilitation; Behavioral: Time-Restricted Eating

INTERVENTIONS:
Behavioral: Standard cardiac rehabilitation — Standard, multi-dimensional cardiac rehabilitation program.
Behavioral: Time-Restricted Eating — Counselling to restrict their eating to between 11 am and 7 pm and to consume water-only for the remaining 16 hours per day
  Arms: Standard cardiac rehabilitation + TRE

SUMMARY:
This study will use a form of intermittent fasting called time-restricted eating (TRE) where individuals consume ad libitum energy intake within a set window of time, commonly 8 hours, which induces a fasting window of 16 hours per day (i.e., 16:8 TRE). TRE could be an effective addition to cardiac rehabilitation as it has demonstrated cardiovascular health benefits and potential for synergy when combined with exercise training. This study will determine if TRE is a feasible and safe nutrition intervention during cardiac rehabilitation and if TRE improves the health benefits of cardiac rehabilitation compared to cardiac rehabilitation alone.

DETAILED DESCRIPTION:
HYPOTHESIS

1. Cardiac rehabilitation and TRE will be feasible in terms of adherence to a 16-hour daily fast (≥70%, which would represent 5/7 days/week) and safe (no excess symptoms or adverse events)
2. Cardiac rehabilitation and TRE will provide added cardiovascular health benefits (improved VO2peak, reduced fat mass) compared to cardiac rehabilitation alone.

JUSTIFICATION: Past animal and human clinical trials have demonstrated TRE to be beneficial in realigning circadian rhythm, improve coronary artery disease (CAD) and peripheral artery disease (PAD) through the reduction in calorie intake, and promote cell signalling and repair pathways during the fasting period. TRE has not been tested in patients with CAD or other heart diseases but has shown to improve comorbid conditions (diabetes and hypertension) and improve metabolic profiles (blood pressure, hemoglobin A1c, fasting glucose, insulin sensitivity, and lipid profiles. Additionally, TRE when combined with exercise, such as in cardiac rehabilitation programs, improves VO2 peak and reduces fat mass compared to exercise alone. The proposed study will deliver a TRE intervention in combination with the cardiac rehabilitation program and is expected to be feasible, safe, and improve outcomes of cardiac rehabilitation.

OBJECTIVES: The primary aim of this study is to evaluate the feasibility (adherence) and safety (adverse events) of TRE in combination with cardiac rehabilitation.

The secondary aim is to assess the efficacy of the intervention on:

1. VO2peak, body composition, fasted glucose, hemoglobin A1c, blood pressure and waist circumference
2. Lifestyle behavioral change outcomes (dietary intake, dietary quality, physical activity, perceived stress)

4.Cardiac rehabilitation adherence

Exploratory aims of the study include identifying sex differences (equal recruitment of males and females) and participants' experience with TRE (including confidence in maintaining this eating pattern or modifications to increase adherence).

RESEARCH METHOD This study will be a two-site (Toronto Rehabilitation Institute and Toronto Western Hospital), 2-arm, parallel-group, randomized feasibility trial of cardiac rehabilitation alone or cardiac rehabilitation plus 16:8 TRE. Men and women who are referred through the standard clinical pathways for coronary artery disease and are willing to accept random assignment and complete the study assessments will be enrolled. Both groups will receive the standard, multi-dimensional cardiac rehabilitation program consisting of physician-directed risk factor management, an individualized exercise prescription, and virtual education. Participants randomized to the TRE group will be asked to eat only between 11 am and 7 pm for the duration of the cardiac rehabilitation program (~16 weeks). Adherence will be collected via twice daily text messages asking participants to respond with the time they started and stopped eating. Safety will be collected by self-report and medical records. Efficacy outcomes will be assessed by cardiopulmonary exercise test, blood draw, dual x-ray absorptiometry, 3-day diet records, accelerometers, and questionnaires. Study outcomes will be measured at baseline and at the end of the cardiac rehabilitation program.

STATISTICAL ANALYSIS Participant characteristics will be summarized using descriptive statistics. For adherence, both the text message response rate and adherence rate to the 16-hour daily fast will be reported. The change in caloric intake, diet quality, physical activity and efficacy outcomes will be compared between groups by analysis of covariance with baseline values as covariates. Relative risk will be used to compare the incidence of safety outcomes between groups. The primary analysis will be intention to treat and performed with both sexes combined. Secondary analyses will be performed separately in each sex.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are referred and eligible for either the outpatient cardiac rehabilitation program for coronary artery disease or peripheral vascular disease
* willing to accept random assignment and complete the study assessments
* Equal numbers of men and women will be recruited

Exclusion Criteria:

* Inability to complete the consent form and communicate in English
* Self-reported history of an eating disorder
* Current or recent (1 year) pregnancy or breast feeding
* Body mass index <18.5 kg/m^2 or clinical signs of cachexia
* Contraindications or inability to perform cardiopulmonary exercise testing
* Type 1 diabetes
* Type 2 diabetes that requires exogenous insulin
* Working night or rotating shifts
* Eating window <12 hours or consistently eating less than 3 meals/day in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to the daily ≥16-hour fast for the 16-weeks of the cardiac rehabilitation program. | Averaged over the 16 weeks of the intervention
  Assessed daily through a custom twice daily automated text message (or email) program, or written logs for those without cell phones. Adherence will be measured as a % of days with ≥16-hour fast.
Cardiorespiratory fitness as measured by peak volume of oxygen consumption (VO2peak) | 16 weeks
  Assessed by an incremental, to-maximum cardiopulmonary treadmill exercise test.
Fat mass | 16 weeks
  Assessed by dual absorptiometry x-ray (DXA) scan.

SECONDARY OUTCOMES:
Symptoms from TRE | 16 weeks
  Self-report of various nutritional impact adverse events collected at support phone calls for both groups
Seattle Angina Questionnaire score | 16 weeks
  Standard scoring of Seattle Angina Questionnaire (minimum = 0, maximum = 100, higher score means better outcome)
Adverse events | 1-year
  re-hospitalizations, recurrent cardiac events, death extracted from medical records
Fat-free mass | 16 weeks
  Assessed by dual absorptiometry x-ray (DXA) scan.
Hemoglobin A1c | 16 weeks
  Measured by blood draw
Blood pressure | 16 weeks
  Systolic and diastolic blood pressure will manually assessed as the average of the 2nd to 6th measurements
Waist circumference | 16 weeks
  Measured by an inelastic tape at the level of the top of iliac crest as the average of two measurements
Fasted blood glucose | 16 weeks
  Measured by fasted blood draw
Metabolic syndrome | 16 weeks
  As defined by the NCEP/ATP III criteria
Lipid profile | 16 weeks
  Individual measures and ratios of total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides from fasted blood draw
Health-related quality of life measured by the RAND-36 Physical Component Summary | 16 weeks
  Physical component summary of the RAND-36 questionnaire (minimum = 0, maximum = 50, higher score is better outcome)

OTHER OUTCOMES:
Macronutrient ratios | 16 weeks
  3-day food record analysed by food analysis software to estimate macronutrient intake
Caloric intake | 16 weeks
  3-day food record analysed by food analysis software to estimate intake
Cardiac rehabilitation adherence | 16 weeks
  The participant's clinical chart for the cardiac rehabilitation program will be reviewed to extract adherence data to the standard components of the program (exercise, nutrition, education, social worker)
Time-restricted eating experience | 16 weeks
  At the end of the intervention, the TRE group will complete a researcher developed questionnaire that asks questions about acceptability of TRE and confidence in continuing the intervention long-term
Mediterranean Diet Score | 16 weeks
  Standard scoring of 14-item Mediterranean Diet Score Tool (minimum = 0, maximum = 14, higher score indicates better outcome)
Physical activity and sedentary time | 16 weeks
  Participants will wear an accelerometer device for 5 days with 3 full days used for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oh, MD, Study Director — University Health Network, Toronto; Amy Kirkham, PhD, Principal Investigator — University of Toronto, KITE Research Institute
Locations (1):
- Toronto Rehabilitation Institute, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No